CLINICAL TRIAL: NCT06980623
Title: Comparative Effectiveness of Tirzepatide vs Semaglutide in Participants With Type 2 Diabetes and Heart Failure With Preserved Ejection Fraction
Status: Active, not recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elisabetta Patorno, MD, DrPH, Brigham and Women's Hospital
Other Study IDs: 2024P001317-2
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Heart Failure
Keywords: Tirzepatide; Semaglutide; Type 2 diabetes; Heart failure; Cardiovascular disease; Mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Cardiovascular Diseases | interventions — Tirzepatide; semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tirzepatide: Patients who initiated tirzepatide with no use in the prior 180 days
  Interventions: Drug: Tirzepatide
- Semaglutide: Patients who initiate semaglutide with no use in the prior 180 days
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Tirzepatide — Exposure group
  Groups: Tirzepatide
Drug: Semaglutide — Referent group
  Groups: Semaglutide

SUMMARY:
This cohort study aims to assess the comparative effectiveness of tirzepatide versus semaglutide with respect to cardiovascular events in patients with type 2 diabetes and heart failure with preserved ejection fraction.

DETAILED DESCRIPTION:
Both semaglutide, a glucagon-like peptide-1 receptor agonist (GLP-1RA), and tirzepatide, a glucose-dependent insulinotropic polypeptide (GIP)/GLP-1RA, are currently approved treatments to control blood glucose in patients with type 2 diabetes (T2D) and to lower weight in patients with obesity, with or without T2D. Obesity is a leading risk factor for the onset and the progression of heart failure (HF), especially HF with preserved ejection fraction (HFpEF). Due to their potent weight-lowering action, semaglutide and tirzepatide have been recently evaluated in placebo-controlled trials conducted among persons with obesity and HFpEF, with or without T2D. These trials showed that semaglutide and tirzepatide reduced HF symptoms and HF events, compared to placebo.

In this new user, active comparator cohort study, the investigators will identify commercially insured adults (aged > 18 years) with T2D and HFpEF who initiated treatment with tirzepatide or semaglutide between June 1, 2022, and December 31, 2024. The investigators will retrieve information for each study participants using deidentified, longitudinal insurance claims data, including demographic characteristics, health plan enrollment status, inpatient and outpatient diagnoses, procedures, health care visits, hospitalizations, and pharmacy dispensing records.

Cohort entry is the day of initiation of tirzepatide or semaglutide. The follow-up starts on the day after cohort entry and continue until the occurrence of an outcome, discontinuation, switching, death, end of continuous health plan enrollment or end of the study period. Our primary outcome is a composite of hospitalization for HF or all-cause mortality.

The investigators will use propensity score adjustment to mitigate the risk of confounding. The investigators will calculate the number of events, incidence rates, and rate differences per 1000 person-years. Cox proportional hazard models will be used to estimate hazard ratios with their 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are new users of tirzepatide or new users of semaglutide
* Patients with diagnosis of T2D and HFpEF, i.e., EF >= 45%.
* Age >= 18 years old
* Patients with continuous health plan enrollment before and including the treatment initiation date

Exclusion Criteria:

* Patients with missing age or sex information
* Patients with type 1 diabetes mellitus, secondary or gestational diabetes
* History of diabetes related complications
* Patients with related chronic diseases.
* History of gastrointestinal conditions.
* Previous exposure to other GLP-1RA and pramlintide
* Patients with prescription dispensing for both tirzepatide and semaglutide on cohort entry date

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients > 18 years old with T2D and HFpEF.
Sampling Method: Non-Probability Sample
Enrollment: 26000 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for heart failure and all-cause mortality | From treatment initiation to end of follow up, up to 48 months.
  Cardiovascular outcome includes hospitalization for HF and all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States